CLINICAL TRIAL: NCT04934514
Title: A Phase I/IIa Study of IAH0968 in Patients With HER2-positive Advanced Solid Tumors
Brief Title: Clinical Study of IAH0968 in Patients With HER2-positive Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SUNHO（China）BioPharmaceutical CO., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IAH0968-I/IIa
Record Dates: First submitted 2021-06-07; First posted 2021-06-22 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-03

CONDITIONS: Advanced Solid Tumor
Keywords: HER2-positive; Advanced Solid Tumor
MeSH Terms: interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ia stage-Dose escalation (Experimental): Using the "3+3" model, 1 subject was included in the 6 mg/kg dose group, and then 3 to 6 patients with HER2-positive advanced solid tumors that failed standard treatment were included in the fixed 3 dose groups (10 mg/kg, 15 mg/kg, and 20 mg/kg) .
  Interventions: Biological: IAH0968
- Ib stage-Dose extension (Experimental): In the three fixed dose groups (10 mg/kg, 15 mg/kg and 20 mg/kg), when a certain dose group meets the condition of increasing the dose to the higher dose (after the DLT observation period for the last subject in the dose group), the second phase of the dose expansion study for this dose group can be carried out. Each dose group includes 6 patients with HER2-positive advanced solid tumors who have failed the standard treatment, and the interval between enrollment is determined by the investigator.
  Interventions: Biological: IAH0968
- IIa stage-Single-agent study (cohort 1) (Experimental): After the completion of the dose escalation in the 20 mg/kg dose group (Phase Ia), a total of 30 patients with HER2-positive advanced biliary system tumors who have failed standard treatment will be enrolled in the 20 mg/kg dose group. Every 3 weeks is a cycle, and the drug is administered once on the first day of each cycle, and the treatment is continued until any end-point event occurs.
  Interventions: Biological: IAH0968
- IIa stage - IAH0968 combined GP regimen study (cohort 2) (Experimental): After the completion of the dose escalation in the 20 mg/kg dose group (phase Ia), a total of 30 patients with newly treated HER2-positive advanced biliary system tumors will be enrolled in the 20 mg/kg dose group combined with the GP regimen (gemcitabine + cisplatin) . Every 3 weeks is a cycle, treatment until any end-point event occurs.
  Interventions: Biological: IAH0968; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Biological: IAH0968 — IAH0968 is an investigational product.
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 intravenous infusion
  Arms: IIa stage - IAH0968 combined GP regimen study (cohort 2)
Drug: Cisplatin — Cisplatin 75 mg/m^2 intravenous infusion
  Arms: IIa stage - IAH0968 combined GP regimen study (cohort 2)

SUMMARY:
This is a phase I/IIa study to evaluate the safety, tolerability and preliminary efficacy of IAH0968 in patients with HER2-positive advanced solid tumors who have failed standard treatment.

DETAILED DESCRIPTION:
The purpose of the Phase Ia/Ib study is to evaluate the tolerability, safety, PK, immunogenicity and preliminary anti-tumor activity of IAH0968 in Chinese subjects. Phase Ia is a dose escalation, and it is planned to recruit about 10-19 subjects with HER2-positive advanced malignancies who have failed standard treatment. Phase Ib is a dose expansion, and it is planned to recruit approximately 18 subjects with HER2-positive advanced malignancies who have failed standard treatment. Phase IIa mainly investigates the effectiveness and safety of IAH0968 in HER2-positive subjects with advanced biliary system tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Phase Ia and Ib: Aged 18 to 65 years old male and female; Phase IIa :Aged 18 to 75 years old male and female
2. Phase I study: Phase Ia and Phase Ib will enroll patients with HER2-positive advanced solid tumors who were confirmed by histopathology and/or cytology and who had failed standard treatments.
3. Phase IIa study: Cohort 1 will enroll patients with HER2-positive advanced biliary system tumors who were confirmed by histopathology and/or cytology and failed standard treatment. Cohort 2 will enroll patients with newly treated HER2-positive advanced biliary system tumors diagnosed by histopathology and/or cytology.
4. According to the RECIST 1.1 standard, at least one measurable lesion exists, and the measurable lesion has not received local treatment (including local radiotherapy, ablation, and interventional therapy).
5. ECOG performance status 0-1.
6. Laboratory examination should meet: ① Blood routine: hemoglobin (HGB) ≥100 g/L, white blood cell count (WBC) ≥3.0×10^9/L, neutrophil count (ANC) ≥1.5×10^9/L, platelet count ( PLT) ≥75×10^9/L; ②Blood biochemistry: total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0×ULN, serum creatinine ( Cr)≤1.5×ULN or calculate the creatinine clearance ≥50 mL/min according to the Cockcroft-Gault formula method.
7. Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiography.
8. Life expectancy ≥3 months.
9. Agree to use at least one medically approved contraceptive method during the trial period and at least 6 months after the last dose (female patients: such as intrauterine devices, contraceptives or condoms, etc.; male patients: such as condoms, abstinence, etc.). Female patients must be non-lactating.
10. Subjects must be fully informed of the content, process and possible risks and benefits of the research and sign the informed consent form. Good compliance, able to complete the study and follow-up.

Exclusion Criteria:

1. Known to have hypersensitivity to any monoclonal antibody.
2. Not recovered from the adverse reactions caused by previous anti-tumor treatments (refer to CTCAE 5.0 to judge, hematological toxicity ≥ 2 grade, non-hematological toxicity ≥ 1 grade). Long-term toxicity after radiotherapy, which is judged to be irreversible by researchers, such as hair loss and pigmentation are excluded.
3. Previously received allogeneic hematopoietic stem cell transplantation or solid organ transplantation.
4. Have undergone surgery within 4 weeks before enrollment, and the investigator believes that the patient's state has not recovered to the point where the study can be started.
5. Received a preventive vaccine or attenuated vaccine or have received blood transfusion within 4 weeks before joining the group.
6. Stage Ia and Stage Ib: Patients who have received trastuzumab and its biosimilar drugs (including single drugs, combination chemotherapy, ADC drugs, bispecific antibodies, etc.) 6 months before enrollment. Stage IIa: Patients who have previously received anti-HER2 therapy.
7. Have received any systemic anti-tumor therapy within 4 weeks before enrollment.
8. Participated in other clinical trials within 4 weeks before enrollment and used clinical research drugs during this period.
9. Central nervous system metastases with clinical symptoms were found within 4 weeks before enrollment. Patients who have previously received treatment for brain or meningeal metastases, if clinical stability has been maintained for at least 2 months, and have stopped systemic hormone therapy (dose>10 mg/day prednisone or other curative hormones) for more than 4 weeks can be included.
10. Patients with ascites (ascites), pleural effusion (pleural effusion) or pericardial effusion that cannot be controlled by drainage or other methods.
11. Past or present suffering from other malignant tumors (except for cured skin basal cell carcinoma and cervical carcinoma in situ).
12. Suffer from serious or poorly controlled diseases, including but not limited to: ① Myocardial infarction, unstable angina pectoris, clinically significant arrhythmias requiring treatment, congestive heart failure, pericarditis, myocarditis, etc. occurred within 6 months before enrollment. ②Hepatitis B virus (HBV) infection and HBV DNA positive (>1×10^3 copies/mL or >500 IU/mL), hepatitis C virus (HCV) infection and HCV RNA positive (>1×10^3 copies/mL or >100 IU/mL), human immunodeficiency virus (HIV) test positive; ③ poorly controlled diabetes, hypertension, thyroid disease, etc.; ④ severe and uncontrollable lung disease (severe infectious pneumonia, interstitial lung disease) Etc.) (≥CTCAE level 3); ⑤Severe infections that cannot be controlled (≥CTCAE level 3).
13. With any situations that the researcher considers inappropriate to participate in this research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) and SAEs (Phase Ⅰ) | 3 months after end event visit
  To investigate the safety characteristics.
Dose limiting toxicities (DLTs) (Phase Ⅰ) | 21 days after first dose
  To determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D).
Objective response rate (ORR) in dose expansion (Phase Ⅱa) | Baseline through up to 2 years or until disease progression
  To explore the clinical effectiveness. Tumor response based on RECIST 1.1.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Cmax (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Cmax) following single dose.
Pharmacokinetic (PK) Cmin (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Cmin) following single dose.
Pharmacokinetic (PK) Tmax (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Tmax) following single dose.
Pharmacokinetic (PK) AUC 0-t (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (AUC 0-t) following single dose.
Pharmacokinetic (PK) AUC 0-∞ (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (AUC 0-∞) following single dose.
Pharmacokinetic (PK) CL (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (CL) following single dose.
Pharmacokinetic (PK) Vd (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Vd) following single dose.
Pharmacokinetic (PK) t1/2 (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (t1/2) following single dose.
Pharmacokinetic (PK) λz (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (λz) following single dose.
Pharmacokinetic (PK) Css,max (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Css,max) following multiple dose.
Pharmacokinetic (PK) Css,min (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Css,min) following multiple dose.
Pharmacokinetic (PK) Css,av (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Css,av) following multiple dose.
Pharmacokinetic (PK) AUCss (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (AUCss) following multiple dose.
Pharmacokinetic (PK) CLss (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (CLss) following multiple dose.
Pharmacokinetic (PK) Vss (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (Vss) following multiple dose.
Pharmacokinetic (PK) R (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (R) following multiple dose.
Pharmacokinetic (PK) DF (Phase Ⅰ) | Day1，2，3，4，6，8，11，14，17，21 of each subsequent cycle (each cycle is 21 days), and at the End of Treatment visit, up to about 2 years
  PK parameters (DF) following multiple dose.
Objective response rate (ORR) in dose escalation (Phase Ⅰ) | Baseline through up to 2 years or until disease progression
  Tumor response based on RECIST 1.1.
Incidence of adverse events (AEs) and SAEs (Phase Ⅰ) | 3 months after end event visit
  To investigate the safety characteristics.
Immunogenicity of IAH0968 (Phase Ⅰ) | 3 months after end event visit
  The frequency of anti-drug antibodies (ADA) against IAH0968.(Phase Ⅰ)
Progression free survival (PFS) (Phase Ⅱa) | Baseline through up to 2 years or until disease progression
  PFS as assessed using RECIST 1.1.
Overall survival (OS) (Phase Ⅱa) | Baseline through up to 2 years or until disease progression
  OS as assessed using RECIST 1.1.
Disease control rate (DCR) (Phase Ⅱa) | Baseline through up to 2 years or until disease progression
  DCR as assessed using RECIST 1.1.
Incidence of adverse events (AEs) and SAEs (Phase Ⅱa) | 3 months after end event visit
  To investigate the safety characteristics.
Immunogenicity of IAH0968 (Phase Ⅱa) | 3 months after end event visit
  The frequency of anti-drug antibodies (ADA) against IAH0968.(Phase Ⅱa)

CONTACTS AND LOCATIONS:
Overall Officials: Yunpeng Liu, MD, Principal Investigator — First Hospital of China Medical University
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song N, Teng Y, Shi J, Teng Z, Jin B, Qu J, Zhang L, Yu P, Zhao L, Wang J, Li A, Tong L, Jiang S, Liu Y, Yin L, Jiang X, Xu T, Cui J, Qu X, Liu Y. A novel anti-HER2 monoclonal antibody IAH0968 in HER2-positive heavily pretreated solid tumors: results from a phase Ia/Ib first-in-human, open-label, single center study. Front Immunol. 2024 Nov 29;15:1481326. doi: 10.3389/fimmu.2024.1481326. eCollection 2024. PMID 39676868